CLINICAL TRIAL: NCT01400269
Title: An Evaluation of a Developmentally-Based Parent Training Program for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-11022010-7169
Record Dates: First submitted 2011-05-31; First posted 2011-07-22 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Autistic Disorder
Keywords: PACE
MeSH Terms: conditions — Autistic Disorder | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pacific Autism Center for Education (PACE) (Experimental): Behavioral: Pacific Autism Center for Education (PACE) developmentally based parent delivered intervention
  Interventions: Behavioral: Pacific Autism Center for Education (PACE ) developmentally based parent delivered intervention

INTERVENTIONS:
Behavioral: Pacific Autism Center for Education (PACE ) developmentally based parent delivered intervention — Pacific Autism Center for Education (PACE ) developmentally based parent delivered intervention

SUMMARY:
The purpose of this study is to assess the efficacy of a parent training program in the treatment of social and communication deficits in children with autism. Specifically, this study will evaluate a developmentally based parent delivered intervention in the community developed by Pacific Autism Center for Education (PACE).

DETAILED DESCRIPTION:
There are many treatments that claim to be effective for children with autism; however many of these treatments have not been investigated using scientifically rigorous methodology. A variety of developmentally based parent delivered interventions are gaining popularity as a type of treatment parents utilize to improve symptoms related to their child's diagnosis of autism. Pacific Autism Center for Education (PACE)is a agency that provides a developmentally based parent delivered intervention in the community. Currently, this parent training program has not been evaluated using scientific methodology. Investigation into this community delivered treatment and its effectiveness to improve social and communication deficits will aid clinicians in providing better care for children with autism.

ELIGIBILITY:
Inclusion Criteria:

* meets DSM-IV-TR criteria for an autism spectrum disorder (pervasive developmental disorder) on the basis of clinical evaluation and the research diagnostic methods
* age range between 18 months and 6.11 years
* male or female in good medical health
* will be starting PACE parent training program
* intends on continuing PACE program for a minimum of 12 weeks

Exclusion Criteria:

* medically unstable (e.g., more than one seizure a month)
* a medical diagnosis that causes autism like symptomology (e.g., Fragile X, Down syndrome, Angelman's syndrome, tuberous sclerosis, Rett's disorder)

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Social Responsiveness Scale | Baseline and Week 12
  Outcome measure is the change from week 12 relative to baseline.

SECONDARY OUTCOMES:
Repetitive Behavior Scale | Baseline and Week 12
  Outcome measure is the change from week 12 relative to baseline.
Family Empowerment Scale | Baseline and Week 12
  Outcome measure is the change from week 12 relative to baseline.
Caregiver Strain questionnaire | Baseline and Week 12
  Outcome measure is the change from week 12 relative to baseline.
Pediatric Quality of Life Inventory | Baseline and Week 12
  Outcome measure is the change from week 12 relative to baseline.
Sensory Profile Questionnaire | Baseline and Week 12
  Outcome measure is the change from week 12 relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Gengoux GW, Schapp S, Burton S, Ardel CM, Libove RA, Baldi G, Berquist KL, Phillips JM, Hardan AY. Effects of a parent-implemented Developmental Reciprocity Treatment Program for children with autism spectrum disorder. Autism. 2019 Apr;23(3):713-725. doi: 10.1177/1362361318775538. Epub 2018 May 18. PMID 29775078